CLINICAL TRIAL: NCT06485544
Title: A Multicenter Randomized Controlled Trial of Neoadjuvant Adebrelimab Combined With Chemotherapy for Resectable Small Cell Lung Cancer (SCLC)
Brief Title: Neoadjuvant Adebrelimab in Resectable SCLC: A Randomized Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT202405-04
Record Dates: First submitted 2024-06-20; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Small Cell Lung Cancer (SCLC)
Keywords: SCLC; Adebrelimab; Neoadjuvant; Chemotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adebrelimab + Etoposide + Platinum-based Therapy (Experimental): Participants in this arm will receive Adebrelimab, Etoposide, and Platinum-based therapy. Adebrelimab will be administered intravenously at a fixed dose of 1200 mg over 30 minutes on Day 1 of each 3-week cycle. Following Adebrelimab, Etoposide will be given at a dose of 100 mg/m2 via intravenous infusion over 30 minutes on Days 1 to 3 of each cycle. Concurrently, Platinum-based therapy (either Cisplatin at AUC5 or Carboplatin at AUC5 or Cisplatin at 100 mg/m2) will be administered via intravenous infusion on Day 1 of each cycle. This treatment regimen will be repeated for 3-4 cycles, with a 4-6 week drug-free interval before surgical treatment.
  Interventions: Drug: Adebrelimab + Etoposide + Platinum-based Therapy
- Etoposide + Platinum-based Therapy (Active Comparator): Participants in this arm will receive Etoposide and Platinum-based therapy. Etoposide will be administered at a dose of 100 mg/m2 via intravenous infusion over 30 minutes on Days 1 to 3 of each 3-week cycle. Concurrently, Platinum-based therapy (either Cisplatin at AUC5 or Carboplatin at AUC5 or Cisplatin at 100 mg/m2) will be administered via intravenous infusion on Day 1 of each cycle. This treatment regimen will be repeated for 3-4 cycles, with a 4-6 week drug-free interval before surgical treatment.
  Interventions: Drug: Etoposide + Platinum-based Therapy

INTERVENTIONS:
Drug: Adebrelimab + Etoposide + Platinum-based Therapy — Intervention Description for Treatment Group:
  This intervention includes Adebrelimab in combination with Etoposide and Platinum-based therapy as neoadjuvant treatment for resectable small cell lung cancer (SCLC). Adebrelimab is administered intravenously at a fixed dose of 1200 mg over 30 minutes on Day 1 of each 3-week cycle, followed by Etoposide at a dose of 100 mg/m2 via intravenous infusion over 30 minutes on Days 1 to 3 of each cycle. Concurrently, Platinum-based therapy (either Cisplatin at AUC5 or Carboplatin at AUC5 or Cisplatin at 100 mg/m2) is administered via intravenous infusion on Day 1 of each cycle. The treatment regimen consists of 3-4 cycles, with a 4-6 week drug-free interval before surgical treatment.
  Arms: Adebrelimab + Etoposide + Platinum-based Therapy
Drug: Etoposide + Platinum-based Therapy — Intervention Description for Control Group:
  This intervention includes Etoposide in combination with Platinum-based therapy as neoadjuvant treatment for resectable small cell lung cancer (SCLC). Etoposide is administered at a dose of 100 mg/m2 via intravenous infusion over 30 minutes on Days 1 to 3 of each 3-week cycle. Concurrently, Platinum-based therapy (either Cisplatin at AUC5 or Carboplatin at AUC5 or Cisplatin at 100 mg/m2) is administered via intravenous infusion on Day 1 of each cycle. The treatment regimen consists of 3-4 cycles, with a 4-6 week drug-free interval before surgical treatment.
  Arms: Etoposide + Platinum-based Therapy

SUMMARY:
This study is a randomized, open-label, multicenter exploratory research aiming to evaluate the efficacy and safety of Adebrelimab in combination with chemotherapy (etoposide and platinum-based therapy) as neoadjuvant treatment for resectable stage I-IIIB (stage IIIB limited to T1-4N1-2M0) small cell lung cancer (SCLC). The study is primarily conducted at Tangdu Hospital of the Fourth Military Medical University. A total of 104 patients with stage IA-IIIB SCLC (stage IIIB limited to T1-4N1-2M0) will be enrolled and randomized 1:1 to receive either Adebrelimab plus chemotherapy or chemotherapy alone. Each patient will undergo 3 cycles of study treatment followed by a 3-4 week break before surgery. Treatment will be discontinued if patients experience disease progression, intolerable drug-related adverse events, withdrawal of informed consent, or other specified conditions during the study. Effectiveness and safety outcomes will be monitored throughout the trial. The primary objective is to evaluate pathological complete response (pCR) with Adebrelimab combination therapy. Secondary objectives include assessing event-free survival (EFS), major pathological response (mPR), objective response rate (ORR), disease-free survival (DFS), and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years, inclusive, with no restriction on gender.
2. ECOG performance status of 0-1.
3. Histologically or cytologically confirmed diagnosis of small cell lung cancer (SCLC).
4. According to the 8th edition of AJCC staging, participants must have resectable or potentially resectable stage I-IIIB (T1-4N0-2M0) SCLC.
5. Measurable lesions (tumor lesions with a CT scan long axis ≥10 mm, lymph node lesions with a CT scan short axis ≥10 mm).
6. Initial diagnosis of small cell lung cancer without prior treatment with radiation, chemotherapy, traditional Chinese medicine, surgery, or targeted therapy.
7. Various imaging examinations including PET-CT, enhanced CT or ultrasound of the chest and abdomen, MRI of the head, and bone scan confirm no metastatic lesions.
8. Participants must have sufficient cardiopulmonary function to tolerate planned lung resection surgery.
9. No contraindications to immune checkpoint inhibitor (ICI) use based on laboratory tests.
10. Normal organ function, as defined by the following criteria:

(1) Hematological criteria (within 14 days without blood transfusion, hematopoietic factors, or correcting medications):

1. ANC ≥ 1.5 × 10^9/L;
2. PLT ≥ 100 × 10^9/L;
3. Hb ≥ 90 g/L; (2) Biochemical criteria:

a. TBIL ≤ 1.5 × ULN; b. ALT, AST ≤ 2.5 × ULN (if abnormal liver function due to liver metastasis, ≤ 5 × ULN); c. Serum creatinine (sCr) ≤ 1.5 × ULN, estimated glomerular filtration rate (eGFR) ≥ 50 mL/min (Cockcroft-Gault formula); (3) Coagulation function: INR ≤ 1.5 × ULN and APTT ≤ 1.5 × ULN. 11. Female participants of childbearing potential must have a negative serum pregnancy test within 3 days before starting study medication and agree to use a medically accepted method of highly effective contraception during the study and for 3 months after the last dose of study drug (e.g., intrauterine device, contraceptive pills, or condoms). Male participants with female partners of childbearing potential must have undergone surgical sterilization or agree to use effective contraception during the study and for 3 months after the last dose of study drug.

12. Participants must voluntarily consent to participate in this study, sign an informed consent form, demonstrate good compliance, and agree to follow-up visits.

Exclusion Criteria:

1. Central nervous system metastasis.
2. History of any active autoimmune disease or autoimmune disease (including but not limited to moderate or severe interstitial lung disease, uveitis, colitis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism [patients controlled by hormone replacement therapy may be included]); patients with vitiligo or childhood asthma completely resolved without adult intervention may be included; patients requiring bronchodilators for medical intervention are excluded.
3. Congenital or acquired immunodeficiency, such as HIV infection, active hepatitis B (HBV DNA ≥ 500 IU/mL), hepatitis C (HCV antibody positive with HCV-RNA above the lower limit of detection by analytical methods), or co-infection of hepatitis B and C, active pulmonary tuberculosis.
4. Use of immunosuppressive drugs within 14 days prior to the first administration of the study drug, excluding nasal and inhaled corticosteroids or physiological doses of systemic steroid hormones (i.e., no more than 10 mg/day of prednisone or its equivalent).
5. Vaccination with live attenuated vaccines within 4 weeks before the first administration or planned during the study period.
6. Any other malignancy within the past 3 years.
7. Evidence of past or present pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-induced pneumonia, or severely impaired lung function.
8. Uncontrolled hypertension.
9. Grade II or higher myocardial ischemia or myocardial infarction, uncontrolled arrhythmias (including QTc interval ≥450 ms for males and ≥470 ms for females). According to NYHA standards, Class III-IV heart failure, or left ventricular ejection fraction (LVEF) < 50% by cardiac ultrasound, myocardial infarction within 6 months before enrollment, NYHA Class II or higher heart failure, uncontrolled angina, uncontrolled severe ventricular arrhythmias, clinically significant pericardial disease, or electrocardiogram (ECG) indicating acute ischemia or active conduction system abnormalities.
10. Severe infection within 4 weeks before the first administration (e.g., requiring intravenous antibiotics, antifungals, or antivirals), or unexplained fever > 38.5°C during screening/first administration.
11. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
12. Pregnant or breastfeeding women; patients of childbearing potential unwilling or unable to use effective contraception.
13. Known allergic reaction, hypersensitivity, or intolerance to SHR-1316, etoposide, cisplatin, or their excipients.
14. Participation in another clinical study or less than 4 weeks since the end (last dose) of a previous clinical study, or less than 5 half-lives of the study drug.
15. Known history of substance abuse, alcohol abuse, or drug addiction.
16. Any condition that the investigator believes may compromise the safety of the participant or the participant's ability to meet or follow study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate(pCR) | 7 days after surgery.
  Pathologic complete response (pCR), defined as the absence of tumor cells in all specimens (ypT0N0) .

SECONDARY OUTCOMES:
Event-free survival (EFS) | Long term follow-up will continue until preoperative progression, postoperative recurrence, or death from any cause at least two years.
  The length of time after primary treatment for a cancer ends that the patient remains free of certain complicationsor events that the treatment was intended toprevent or delay.
Major pathologic response (MPR) | 7 days after surgery.
  MPR is defned as less than 10% residual viable tumor after neoadjuvant therapy.
Objective response rate (ORR) | 7 days before surgery
  Per Response Evaluation Criteria in Solid Tumorsersion 1.1(REClST 1.1) using Investigator assessments, is defneas the number (%) of patients with responseof Complete Response or Partial Response.
Disease-free survival(DFS) | Long term follow-up will continue until the death of the subiect or the end of the studv. at least two years
  The length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of that cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital Affiliated to the Fourth Military Medical University, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No